CLINICAL TRIAL: NCT04677413
Title: Phase I Trial of Ultra-fractionated Adaptive Radiotherapy, Chemotherapy and Selective Omission of Surgery for Locally Advanced Rectal Cancer
Brief Title: Ultra-fractionated Radiotherapy for Rectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Nina Sanford, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1394
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer,T3-4 or N+
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective dose evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I Dose Cohorts (Experimental): DOSE LEVEL 1 : 30 Gy (tumor)/ 25 Gy (pelvis)
  DOSE LEVEL 2 : 35 Gy (tumor)/ 25 Gy (pelvis)
  DOSE LEVEL 3 : 40 Gy (tumor)/ 25 Gy (pelvis)
  Interventions: Radiation: Ultrafractionated radiotherapy for rectal cancer

INTERVENTIONS:
Radiation: Ultrafractionated radiotherapy for rectal cancer — To determine the toxicity of dose-escalated hypofractionated RT, in patients with locally advanced rectal cancer treated with RT, FOLFOX or CAPOX chemotherapy and selective omission of surgery.

SUMMARY:
The rationale of this clinical trial is to assess the feasibility of selective non-operative management for locally advanced rectal cancer using dose-escalated ultra-fractionated short course radiation therapy interdigitated with chemotherapy. We believe delivering short course radiotherapy over a prolonged interval, at escalated doses and with concurrent chemotherapy may be feasible and allow for improved clinical response.

DETAILED DESCRIPTION:
To determine the maximal tolerated dose (MTD) of dose-escalated hypofractionated adaptive RT, in patients with locally advanced rectal cancer treated with RT, FOLFOX (5-FU, oxaliplatin, leucovorin) or CAPOX (capecitabine, oxaliplatin) chemotherapy and selective omission of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age. Both men and women and members of all races and ethnic groups will be included.
2. Willing and able to provide written informed consent
3. Pathologic diagnosis of rectal adenocarcinoma
4. T3-4 and/or N+ disease per AJCC 8th edition
5. No prior treatment for rectal adenocarcinoma
6. Eastern Cooperative Group (ECOG) performance status of 0-2.
7. Laboratory values supporting acceptable organ and marrow function within 30 days of eligibility confirmation. Defined as follows:

   * WBC ≥ 3,000/mL;
   * ANC WBC ≥ 1,000/mL;
   * PLT ≥ 75,000/mL;
   * T Bili ≤ 1.5 x upper limit of normal (ULN);
   * AST/ALT ≤ 2.5 x ULN;
   * Creatinine not above ULN, or creatinine clearance >50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.
8. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) starting with the first dose of study therapy through 90 days after the last dose of study drugs. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Distant nodal disease (retroperitoneal nodes) including inguinal nodes, or any metastatic disease by CT.
2. Prior RT to the pelvis.
3. Uncontrolled comorbid illness or condition including congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric illness that would limit compliance with the study requirements.
4. Psychiatric illness/social situations that would limit consenting and compliance with study requirements.
5. Participants who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose (MTD) of dose-escalated hypofractionated RT. | 0 to 60 days post radiation therapy
  The MTD will be based upon toxicity, which will be assessed according to the NCI's CTCAE v5.0 toxicity criteria. Dose limiting toxicities will include any of the following Grade 3+ GI toxicities.

SECONDARY OUTCOMES:
To evaluate the rate of clinical complete and near complete response to radiation and chemotherapy. | 1 year
  Clinical complete response, assessed at 4-8 weeks after completion of chemotherapy and radiation, will be defined based upon endoscopy and MRI as described in section 4.1.1.
To determine the organ preservation rate at 1 year after radiotherapy and FOLFOX or CAPOX chemotherapy. | 1 year
  Organ preservation rate will be defined as rate of intact rectum and no local regional failure at 1 year from completion of treatment.
To evaluate local regional recurrence, defined as the time between date of therapy initiation and date of local progression. | 1 year
  The rate of local regional recurrence will be defined as disease recurrence in the pelvis and will be recorded on a time interval since completion of treatment. This will be evaluated as a median and rate up to 1 year post treatment. The time will be backdated to when the recurrence was observed.
To evaluate disease-free survival (DFS), defined as the time between date of therapy completion the first date of documented disease progression or death. | 1 year
  The disease-free survival endpoint will be defined as the percent of patients without disease recurrence at 1-year.
For patients undergoing surgery, to evaluate the rate of R0 resection, defined as a negative surgical margin at time of total mesorectal excision. | 1 year
  R0 resection will be defined by the percent of patients with an R0 resection or negative surgical margin at the time of total mesorectal excision. Acute and late toxicities will be recorded as the rate of treatment related grade 3-5 adverse events experienced in the acute phase from initiation of therapy to 6 weeks treatment to the late phase 6 weeks to 1 year, using the NCI's CTCAE v5.0 toxicity criteria.
To evaluate the rate of distant failure, defined as development of disease outside of the pelvis. | 1 year
  The rate of distant failure will be recurrence of disease outside of the pelvis that will be collected on time interval since completion of therapy and be evaluated as a median or rate up to 1-year follow-up. Time will be backdated to when the recurrence was observed.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Sanford, MD, Principal Investigator — UT SOUTHWESTERN medical CENTRE
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No